CLINICAL TRIAL: NCT07181005
Title: Application of the Validity and Reliability of the Enhanced Paper Grasping Test in Patients With Stroke
Brief Title: The Validity and Reliability of an Improved Paper Grasping Test for Stroke
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Physiotherapy and Rehabilitation Department, Assistant Professor, Sanko University
Other Study IDs: hakanpolat5
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Balance; Validity and Safety
Keywords: stroke; balance; validity and safety
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study included volunteer patients diagnosed with stroke who applied to the Neurology Outpatient Clinic at SANKO University Sani Konukoğlu Application and Research Hospital.

Patients who met the inclusion criteria were evaluated by Dr Hakan Polat and Physiotherapist Fatma Yılmaz in the application laboratory of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, SANKO University.

The assessment form prepared by the researchers will be completed face-to-face with the patients. First, the individuals' demographic information and disease information (how many years ago they were diagnosed with stroke, affected side, affected limb, etc.) will be recorded. The mini best test will be used to assess balance and gait. The muscle strength of the plantar flexor muscle groups in the ankle will be assessed using a manual muscle testing device, and quality of life will be assessed using the Stroke-Specific Quality of Life Scale (SSQOL).

As fall problems in patients may be related to balance problems, lower limb muscle weakness, particularly in the ankle, and reduced quality of life, these parameters will also be evaluated. Therefore, in our study, while examining the validity and reliability of the modified paper grip test in individuals with stroke, its correlation with these parameters will also be examined.

Before the tests are administered, the individuals will be given a practical explanation of how the tests are performed. The individuals will be allowed to rest before the assessments. In the tests, the paper grip test will first be administered by Dr Hakan Polat, followed by the mini best test, the assessment of the strength of the ankle plantar and dorsiflexor muscles, and the assessment of quality of life. One week after the applications, only the paper grip test will be re-administered by Fzt. Fatma Yılmaz in the same environment. The individuals in this study will be assessed in the same environment in both sessions. In this way, the effect of environmental factors on the patients' performance will be minimised.

DETAILED DESCRIPTION:
Stroke is one of the most significant diseases causing death and disability worldwide. Stroke is a disease that leads to neurological disorders as a result of the sudden interruption of blood flow in the vessels supplying the brain. It is divided into haemorrhagic and ischaemic stroke. Symptoms vary depending on the affected area of the brain. Common symptoms observed in stroke patients include muscle weakness, reduced upper limb function, difficulty walking, balance and coordination problems, and communication problems.

Stroke patients are at high risk of falling, particularly due to balance problems. Consequently, fear of falling in stroke patients leads to kinesiophobia (fear of movement) and decreases in activities of daily living and difficulties in adaptation.

Balance problems are primary abnormal motor characteristics in individuals who have had a stroke, and it has been shown that they are the primary problem in approximately 80% of cases, leading to walking disorders, posture disorders, and falling problems.

Based on this information, balance rehabilitation must be a primary focus in stroke rehabilitation for falling problems. A detailed balance assessment is of great importance for rehabilitation treatment. According to research in the literature, balance assessment in individuals who have suffered a stroke is generally performed statically and dynamically. The functional reach test, functional balance scale, and timed up and go test are generally preferred. However, it is thought that the main source of balance problems is lower extremity muscle strength loss. Although there is a significant relationship between lower extremity muscle strength loss and increased risk of falling in individuals with stroke, current assessment tools do not include direct quantitative assessment, which may weaken their effectiveness.

The Enhanced Paper Grip Test (EPGT) can fill this gap in the literature. The EPGT offers a simple measurement using hallux plantar flexion strength, without the need for special devices or equipment.

The Enhanced Paper Grip Test (EPGT) can be used to assess the risk of falling in individuals with stroke.

It has been suggested that it could be a useful screening tool for assessing the risk of falling in geriatric individuals. The validity and reliability of this test have also been established in individuals diagnosed with multiple sclerosis.

The EPGT is a test that can be performed without requiring a large space, is easy to administer, low-cost, and quick. Therefore, it is an easily applicable test. We aimed to apply it by testing the validity and reliability of the paper grasp test in stroke patients.

Volunteer patients diagnosed with stroke who applied to the SANKO University Sani Konukoğlu Application and Research Hospital Neurology Polyclinic will be included in the study. Patients who meet the inclusion criteria will be evaluated by Dr Hakan Polat and Physiotherapist Fatma Yılmaz in the application laboratory of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, SANKO University. The roles of Associate Professor Zekiye İpek Kırmacı in the study are: planning the study, formulating hypotheses, interpreting the results, and converting them into an article.

The assessment form prepared by the researchers will be completed face-to-face with the patients. First, the individuals' demographic information and disease information (how many years ago they were diagnosed with stroke, affected side, affected limb, etc.) will be recorded. The mini best test will be used to assess balance and gait. The muscle strength of the plantar flexor muscle groups in the ankle will be assessed using a manual muscle testing device, and quality of life will be assessed using the Stroke-Specific Quality of Life Scale (SSQOL).

As fall problems in patients may be related to balance problems, lower limb muscle weakness, particularly in the ankle, and reduced quality of life, these parameters will also be evaluated. Therefore, in our study, while examining the validity and reliability of the modified paper grip test in individuals with stroke, its correlation with these parameters will also be examined.

Before the tests are administered, the individuals will be given a practical explanation of how the tests are performed. The individuals will be allowed to rest before the assessments. In the tests, the paper grip test will first be administered by Dr Hakan Polat, followed by the mini best test, the assessment of the strength of the ankle plantar and dorsiflexor muscles, and the assessment of quality of life. One week after the applications, only the paper grip test will be re-administered by Fzt. Fatma Yılmaz in the same environment. The individuals in this study will be assessed in the same environment in both sessions. In this way, the effect of environmental factors on the patients' performance will be minimised.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-65 with a diagnosis of ischaemic or haemorrhagic stroke
* Voluntarily participating in the study

Exclusion Criteria:

* -Pregnant or within the first 3 months after giving birth
* Anyone who has taken any medication that affects their ability to walk or who has suffered an orthopaedic injury within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Neurology Outpatient Clinic of SANKO University Sani Konukoğlu Application and Research Hospital with a diagnosis of stroke
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Mini Best Test | 1 years
  This is one of the clinical tests used to assess walking and balance. It consists of four sub-parameters: preparatory movement, reactive postural control, sensory orientation, and dynamic walking, comprising a total of 14 items. It is a test scored out of a total of 28 points, taking an average of 10-15 minutes to complete. A high score indicates high function.
Manual muscle testing device | 1 years
  muscle strength (right foot dorsiflexion, left foot dorsiflexion, right foot plantar flexion, left foot plantar flexion) will be measured using the Commander Echo brand manual muscle testing device. The participant will be a
Enhanced Paper Grasping Test | 1 years
  During measurement, participants will sit in a calm environment on a chair without armrests, with their feet and knees at a 90-degree angle, and their upper limbs comfortably placed alongside their torso. This test involves

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko Unıversıty, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be decided when the study is completed